CLINICAL TRIAL: NCT03701295
Title: A Phase Ib/II Study of the Histone Methyltransferase Inhibitor Pinometostat in Combination With Azacitidine in Patients With 11q23-Rearranged Acute Myeloid Leukemia
Brief Title: Pinometostat and Azacitidine in Treating Patients With Relapsed, Refractory, or Newly Diagnosed Acute Myeloid Leukemia With 11q23 Rearrangement
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02128; NCI-2018-02128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10200 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10200 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia With t(9;11)(p21.3;q23.3); MLLT3-MLL; Leukemia Cutis; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; EPZ-5676

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pinometostat, azacitidine) (Experimental): Patients receive pinometostat IV continuously on days 1-28 and azacitidine IV over 10-40 minutes or SC for 7 of the first 10 days of the cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Pinometostat

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Pinometostat — Given IV
  Other Names: DOT1L Inhibitor EPZ-5676; EPZ-5676

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of pinometostat when given together with azacitidine and to see how well it works in treating patients with acute myeloid leukemia that has come back (relapsed), does not respond to treatment (refractory), or is newly diagnosed, with an 11q23 rearrangement. Pinometostat and azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the combination of pinometostat, at a dose of 54 or 90 mg/m^2/day, and azacitidine, at a dose of 75 mg/m^2 daily for 7 days, is safe and tolerable in patients with MLL-rearranged acute myeloid leukemia, either in the relapsed/ refractory setting or in those who choose not to undergo standard induction therapy in the previously untreated setting. (Phase Ib) II. To determine the preliminary efficacy, as determined by overall response rate (complete response [CR], complete response with incomplete bone marrow recovery [CRi], partial response [PR], and morphologic leukemia-free state [MLFS]), of pinometostat administered at the maximum tolerated dose from the phase 1b, combined with azacitidine administered at 75 mg/m^2 daily for 7 days, in patients with MLL-rearranged acute myeloid leukemia, either in the relapsed/refractory setting or in those who choose not to undergo standard induction therapy in the previously untreated setting. (Phase II)

SECONDARY OBJECTIVES:

I. Perform correlative studies to evaluate for on-target effects, cellular differentiation, and decreased leukemia cell proliferation in these patients. (Phase Ib and II) II. To observe and record anti-tumor activity. (Phase Ib)

OUTLINE: This is a phase Ib, dose-escalation study of pinometostat followed by a phase II study.

Patients receive pinometostat intravenously (IV) continuously on days 1-28 and azacitidine IV over 10-40 minutes or subcutaneously (SC) for 7 of the first 10 days of the cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed acute myeloid leukemia
* Patients must have an 11q23 translocation or partial tandem duplication, confirmed by cytogenetics, fluorescence in situ hybridization (FISH), or myeloid panel. Both de novo and therapy-related acute myeloid leukemia (AML) with an 11q23 rearrangement or partial tandem duplication (PTD) are considered eligible
* Patients may not have any other targetable mutations (such as FLT3, IDH1, and IDH2) identified on myeloid mutational panel testing or must refuse treatment with a targeted agent if such a mutation is detected
* Eastern Cooperative Oncology Group (ECOG) performance status < 3 (Karnofsky > 60%)
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x upper limit of normal (ULN)
* Total bilirubin < 2 times the upper limit of institutional normal (ULN) unless due to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 2 times the upper limit of institutional normal (ULN) OR creatinine clearance glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2
* Patients treated in the up-front setting must decline standard-of-care therapy
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity with a close legal guardian/caregiver may be considered
* Patients must have measurable disease, defined as abnormal blasts detectable in the peripheral blood or bone marrow or the presence of extramedullary disease, including leukemia cutis. Patients with extramedullary disease but no bone marrow disease are still considered eligible
* Patients may have had previous treatment with standard-of-care or experimental agents. Patients who have previously undergone bone marrow transplantation may also be included
* Patients who are human immunodeficiency virus (HIV) positive (+), hepatitis B virus (HBV)+, and/or hepatitis C virus (HCV)+ may be eligible as follows:

  * Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial. The antiretroviral therapy should not strongly induce or inhibit CYP3A4
  * If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
  * If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load
* The effects of pinometostat on the developing human fetus are unknown. For this reason and because histone methyltransferase inhibitors as well as hypomethylating agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and for the duration of study participation and for 4 weeks after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of pinometostat and azacitidine administration

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with active central nervous system (CNS) disease are excluded from this clinical trial because they may develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a prior history of CNS disease will not be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pinometostat or azacitidine
* Patients receiving any medications or substances that are inhibitors or inducers of the CYP3A4 or CYP450 system should have their medications reviewed and adjusted for interactions as appropriate for local institutional practice. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients receiving any medications or substances that are inhibitors or inducers of MATE1 and MATE2-K transporters should have their medications reviewed and adjusted for interactions as appropriate for local institutional practice. Pinometostat has been demonstrated to be an inhibitor of MATE1 and MATE2-K transporters in vitro, although the clinical significance of this is unclear. Drug interactions may occur between pinometostat and other therapies that are MATE substrates, including metformin. Consultation with a frequently updated medical reference and/or pharmacist should be sought to guide necessary changes in the patient's other medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled or clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients with these conditions that are medically well controlled may be considered for enrollment
* Pregnant women are excluded from this study because pinometostat is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pinometostat, breastfeeding should be discontinued if the mother is treated with pinometostat. These potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy should have their regimen reviewed for potential pharmacokinetic interactions with pinometostat and azacitidine. In the event of a potential interaction, alternative therapies may be considered in consultation with the patient's primary HIV physician
* Absence of an 11q23 rearrangement or absence of an 11q23 partial tandem duplication
* Patients with an active bleeding diathesis
* Patients at increased risk of QT prolongation (e.g. from known long-QT syndrome) or who have a corrected QT interval that is persistently longer than 450 ms despite adjustments to other medications
* Patients who are eligible for or willing to receive intensive induction therapy for de novo AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Menghrajani, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pinometostat, Azacitidine)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 22 [22 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) (Phase Ib)
Description: Safety and tolerability will be assessed by evaluating the number of patients out of 6 who experience a DLT defined as a significant suspected adverse reaction or clinically significant abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications.
Time Frame: Up to day 42
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate (Phase II)
Description: Will be defined by the 2017 European Leukemia Network guidelines and as the number of patients who achieve a complete response (CR), complete response with incomplete bone marrow recovery (CRi), partial response (PR), or morphologic leukemia-free state (MLFS), with or without minimal residual disease (MRD), at any time point.
Time Frame: Up to the time of count recovery after 6 cycles of combination therapy
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Who Experience a DLT (Phase Ib)
Time Frame: Up to day 42
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in H3K79 Methylation (Phase Ib)
Description: Will compare quantitative methylation and methylation valence (e.g. if H3K27 has been methylated once, twice, or three times) from baseline and subsequent bone marrow samples using descriptive statistics and graphical displays. A Wilcoxon signed rank test will be used to assess post-treatment differences as compared to baseline.
Time Frame: Baseline up to day 28
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Expression Levels of HOXA9 and Meis1 (Phase Ib)
Description: Will compare expression level by quantitative polymerase chain reaction (qPCR) of HOXA9 and Meis1 levels from baseline and subsequent bone marrow samples using descriptive statistics and graphical displays. A Wilcoxon signed rank test will be used to assess post-treatment differences as compared to baseline.
Time Frame: Baseline up to day 28
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

6. Secondary Outcome: Fraction of Cells With 11q23 Rearrangements (Phase Ib)
Description: Samples will be banked, and cytogenetic and fluorescence in situ hybridization (FISH) analysis of these cells will be performed to evaluate for the presence of MLL-rearrangement in patients who respond to therapy.
Time Frame: Up to day 28
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Absolute Neutrophil/Absolute Monocyte Count (Phase Ib)
Description: Will evaluate differentiation by performing a differential on the bone marrow biopsy and peripheral blood samples at baseline and from subsequent time points and assessing percentage of monocytes / neutrophils, bands, and myeloid forms present.
Time Frame: Baseline up to day 28
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Patients Who Experience a DLT (Phase II)
Time Frame: Up to 1 month post-treatment
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

9. Secondary Outcome: Response Rate Based on Relapsed / Refractory or Previously Untreated Status (Phase II)
Description: Patients will be stratified based on treatment for relapsed / refractory or previously untreated disease. The response of each stratum to combination therapy, defined as CR, CRi, MLFS, or PR, with or without MRD, on bone marrow biopsy as defined by the 2017 European Leukemia Network guidelines, will be described. Kaplan-Meier estimates will be calculated and compared for each stratum. A report will be generated to look at all patients, all eligible patients who were enrolled, and all evaluable patients.
Time Frame: Up to 1 month post-treatment
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in H3K79 Methylation (Phase II)
Description: as for outcome 4
Time Frame: Baseline up to 1 month post-treatment
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Expression Levels of HOXA9 and Meis1 (Phase II)
Description: Will compare expression level by qPCR of HOXA9 and Meis1 levels from baseline and subsequent bone marrow samples using descriptive statistics and graphical displays. A Wilcoxon signed rank test will be used to assess post-treatment differences as compared to baseline.
Time Frame: Baseline up to 1 month post-treatment
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

12. Secondary Outcome: Fraction of Cells With 11q23 Rearrangements (Phase II)
Description: Samples will be banked, and cytogenetic and FISH analysis of these cells will be performed to evaluate for the presence of MLL-rearrangement in patients who respond to therapy.
Time Frame: Up to 1 month post-treatment
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Absolute Neutrophil / Absolute Monocyte Count (Phase II)
Description: as for outcome 7
Time Frame: Baseline up to the end of course 1
Population: Did not open Phase 2.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Incorporation of 5-aza-2'-Deoxycytidine Into Genomic Deoxyribonucleic Acid (DNA) and the Extent of Global DNA Methylation (Phase Ib and II)
Description: Will correlate with systemic azacitidine exposure and pharmacodynamics effects.
Time Frame: Up to 1 month post-treatment
Population: Insufficient accrual to analyze this outcome.
Arm/Group | Treatment (Pinometostat, Azacitidine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of study drug.
Arm/Group | Treatment (Pinometostat, Azacitidine)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03701295/Prot_SAP_000.pdf